CLINICAL TRIAL: NCT04597580
Title: Personalised Disease Monitoring During Treatment With an Aromatase Inhibitor + Cyclin Dependent Kinase (CDK) 4/6 Inhibitor as 1st Line Endocrine Therapy in Patients With ER-positive/HER2-negative Metastatic Breast Cancer
Brief Title: Personalised Disease Monitoring in Metastatic Breast Cancer
Acronym: PDM-MBC
Status: Active, not recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTFSp161
Record Dates: First submitted 2019-07-08; First posted 2020-10-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Metastatic; Estrogen Receptor-positive Breast Cancer
Keywords: Breast Neoplasms; Neoplasm Metastasis; Precision Medicine; disease monitoring; Biomarkers, Tumor; Circulating Tumor DNA; Thymidine Kinase
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archived tumour tissue will be analysed using mutation panels to make personalised assays for circulating tumour DNA (dtDNA). ctDNA will be serially collected for subsequent analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with metastatic breast cancer may respond well to treatment and metastases can remain stable for several years. Despite personalised medicine being increasingly used for diagnosis and treatment, follow-up still include radiological response evaluation every 3-4 months, which renders a significant number of 'unnecessary' exams for patients with long-term stable disease. Increasing evidence indicates that tumour markers such as circulating tumour DNA (ctDNA), thymidine kinase 1 (TK1) and cancer antigen 15-3 (CA15-3) may be useful for disease monitoring in the metastatic setting. However, algorithms that accurately define the time-points at which imaging can be foregone or reinstituted when progression is forecast, have not been developed. This study will measure ctDNA, TK1 and CA15-3 at all imaging time-points. The primary aim is to develop an algorithm based on these biomarkers, alone or in combination, that with sufficient specificity and sensitivity can advise whether a scan can be safely omitted at a specific time-point, for patients with MBC receiving first line therapy with AI plus cyclin dependent kinase 4/6 inhibitor (CDK4/6i). Additional samples will be stored such that novel biomarkers can also be tested in future. The cost-effectiveness of using the devised biomarker protocol will be evaluated.

DETAILED DESCRIPTION:
One hundred patients with estrogen receptor positive (ER+)/ Human epidermal growth factor receptor negative (HER2-) metastatic or locally advanced breast cancer, eligible for 1st line endocrine therapy with AI + CDK4/6i will be included. Patients will receive standard therapy (AI + CDK4/6i) and follow-up will proceed according to local guidelines, namely cross sectional imaging with CT thorax/abdomen/pelvis +/- MRI as required and analysis of CA 15-3, every 3 cycles for the first year and every 3-4 cycles thereafter. Participation in the study will include serial blood sampling for the bespoke study biomarkers. Decisions on progression will be made according to the routine imaging tests and the biomarkers will be subsequently analysed.

The investigators hypothesise that the biomarkers ctDNA, TK1 and CA15-3, alone or in combination, will accurately correlate with disease status in patients receiving AI + CDK4/6i for metastatic breast cancer such that routine imaging can be delayed until predefined levels of biomarker progression.

Primary aim: To develop a biomarker-based prediction model to be used in patients with metastatic breast cancer, receiving first line therapy with AI and CDK4/6i, that provides the physician with a recommendation whether or not a radiological examination is required, based on the likelihood that the scan will actually show progressive disease.

Secondary aims

* To define the lead time between rising biomarker and subsequent progression on imaging
* To define the clinical utility of the bespoke biomarkers for disease monitoring
* The relative value of analysing TK1 "on CDK4/6i treatment" versus "off CDK4/6i treatment" for disease monitoring
* To define the economic impact of implementation of the chosen prediction model

ELIGIBILITY:
Inclusion Criteria:

* Confirmed metastatic breast cancer (stage 4) or locally advanced disease not amendable to curative resection. Patients who have locoregional disease only an in whom a response to therapy would lead to potentially curative resection are not eligible.
* ER+/HER2- breast cancer (assessed locally). NOTE: If immunohistochemical analysis is not available from metastatic tissue, the ER and HER2 status from the primary tumour should be used.
* For patients who have had a prior non-breast malignancy within the last 5 years (excluding in situ carcinoma of the cervix and basal cell carcinoma of the skin) biopsy of a metastatic site is required to confirm the diagnosis of metastatic ER+/HER2- breast cancer.
* Eligible for 1st line endocrine treatment with AI + CDK4/6-inhibitor according to local guidelines.

NOTE: ≥ 12 month since termination of adjuvant AI if used NOTE: Patients may have received one prior line of chemotherapy for metastatic breast cancer but should have disease progression at study entry.

* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2 (Oken 1982).
* Life expectancy >3 months.
* Age ≥ 18 years
* Metastatic disease must be radiologically assessable, by means of at least one of the following techniques: computerised tomography (CT) and/or magnetic resonance imaging (MRI), i.e. lesions can be measurable or non-measurable according to RECIST 1.1, but must be clearly evaluable according to the radiologist and/or treating physician. Patients with bone predominant disease who lack evaluable disease on CT according to RECIST 1.1.

must have serial MRI including the representative area in addition to CT TAP. NOTE: Previously irradiated lesions are deemed measurable only if progression is documented at the site after completion of radiation.

- Willing and able to provide informed consent to undergo all trial procedures.

Exclusion Criteria:

* Known CNS metastases, carcinomatous meningitis or leptomeningeal disease unless treated with radiotherapy and symptomatically stable at least 2 weeks after discontinuation of steroids. For such patients, ongoing monitoring of CNS disease is required as standard of care. No screening is needed for asymptomatic patients.
* Concurrent disease(s) or familial, sociological or geographical condition that would, in the investigator's opinion, preclude compliance with study procedures.
* Any serious medical disorder that would compromise the patient's safety.
* Dementia altered mental status, or any psychiatric condition that would prevent the understanding or rendering of Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ER+/HER2- metastatic or locally advanced breast cancer, not amendable for curative surgery, eligible for 1st line endocrine therapy with aromatase inhibitor (AI) + CDK4/6-inhibitor (CDK4/6i).
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood levels of ctDNA, CA15-3 and TK-1 assays from baseline to disease progression | 3-5 years
  ctDNA, CA15-3 and TK-1 assays will be performed at baseline, 2 weeks and at every imaging timepoint to develop a statistical algorithm to predict disease progression that can be tested prospectively in future studies.

SECONDARY OUTCOMES:
Best time for TK1 analysis during CDK4/6i treatment ("on treatment" vs "off treatment") | 3-5 years
  The relative value of analysing TK1 "on CDK4/6i treatment" versus "off CDK4/6i treatment" for disease monitoring

OTHER OUTCOMES:
The economic impact of implementation of the chosen prediction model | 3-5 years
  Cost effectiveness analysis of using the prediction model

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sacha Howell, MD, PhD, Principal Investigator — University of Manchester and The Christie NHS Foundation Trust; Maria Ekholm, MD, PhD, Principal Investigator — University of Gothenburg and Region Jönköping
Locations (7):
- Sweden (5):
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Department of Oncology, Ryhov Hospital, Jönköping
  - Department of Oncology, Kalmar Hospital, Kalmar
  - Department of Oncology, Linköping University Hospital, Linköping
  - Department of Oncology, Södersjukhuset, Stockholm
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Wigan Infirmary, Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mouhanna P, Stahlberg A, Andersson D, Albu-Kareem A, Elinder E, Eriksson O, Kavanagh A, Kovacs A, Larsson KF, Linderholm B, Uminska M, Osterlund T, Howell SJ, Ekholm M. Integration of personalised ultrasensitive ctDNA monitoring of patients with metastatic breast cancer to reduce imaging requirements. Int J Cancer. 2025 Apr 15;156(8):1509-1517. doi: 10.1002/ijc.35292. Epub 2024 Dec 18. PMID 39692755
- [Derived] Brown NL, Howell SJ, Papantoniou D, Eriksson O, Bergqvist M, Williams A, Kavanagh A, Backlund A, Albu-Kareem A, Elinder E, Larsson K, Uminska M, Ekholm M. Prognostic performance of thymidine kinase 1 activity in patients with hormone receptor-positive and HER2-negative metastatic breast cancer treated with CDK4/6 and aromatase inhibitors. Breast Cancer Res Treat. 2026 Feb 11;216(1):6. doi: 10.1007/s10549-025-07879-0. PMID 41670750